CLINICAL TRIAL: NCT05211037
Title: Screening for Renal Complications in Children and Young Adults With Major Sickle Cell Disease
Acronym: NEPHRO-DREPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-AOI-09
Record Dates: First submitted 2022-01-06; First posted 2022-01-27 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Anemia; Sickle Cell Disease
Keywords: Sickle cell disease; Renal complication
MeSH Terms: conditions — Anemia; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kidney function assessment (Experimental)
  Interventions: Diagnostic Test: Kidney function assessment

INTERVENTIONS:
Diagnostic Test: Kidney function assessment — kidney clearance measured by scintigraphy

SUMMARY:
Sickle cell disease is the subject of targeted neonatal screening (carried out when one of the two parents is from an endemic country - sub-Saharan Africa, South-East Asia, Central America, the Caribbean) during the Guthrie test. Haemolysis, which results from the abnormality of the haemoglobin, and the vascular activation it causes, are responsible for multiple organ damage. Major sickle cell syndromes (MSC), by several mechanisms, are responsible for a wide range of renal damage, culminating in end-stage renal failure at an average age of 45 years and with an average survival of 3 years beyond ESRD.

The various renal disorders are : glomerular hyperfiltration and then glomerulosclerosis; tubular dysfunction, especially proximal and distal hyposthenuria (a factor in enuresis); papillary necrosis, renal infarction, episodes of acute renal failure during vaso-occlusive crises; dysregulation of the renin-angiotensin system with early arterial hypertension and, more rarely, extra-membranous glomerulonephritis. In the early stages of these conditions, simple paraclinical tests can identify them before the appearance of specific clinical signs.

In patients suffering from MDS, the HAS (High Authority of Health) recommends an annual check-up carried out in a Competence Centre. According to the HAS recommendations for annual surveillance, in addition to the search for other organic complications, for renal pathology, only microalbuminuria and renal ultrasound are recommended. However, as the literature shows, microalbuminuria and ultrasound only detect some of these renal disorders and at a very late stage. A large number of publications in adults and, to a lesser degree, in children, demonstrate the correlation between the frequency of acute complications of sickle cell disease (episodes of haemolysis, etc.) and the occurrence of kidney damage.

ELIGIBILITY:
Inclusion Criteria:

- Patient over 1 year old followed up in the Competence Centre at the Nice University Hospital, treated for a major sickle cell disease during the annual check-up

Exclusion Criteria:

* Pregnant patients (positive urine pregnancy test)
* Patients with other chronic conditions
* Progressive cancer or kidney disease
* Patients who are breastfeeding

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
renal clearance | at baseline
  renal clearance measured by scintigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Julie BERNARDOR, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No